CLINICAL TRIAL: NCT02540213
Title: Observational Study of MIRCERA in Users of Self-Application and Multidose Systems
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21387
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-11

CONDITIONS: Renal Anemia of Chronic Kidney Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- MIRCERA Ready-To-Use-Syringe: Participants will use MIRCERA ready-to-use-syringes (methoxy polyethylene glycol epoetin beta 0.6 micrograms per kilogram [mcg/kg]) every 2 weeks (q2w) up to 9 months
  Interventions: Device: MIRCERA

INTERVENTIONS:
Device: MIRCERA — Methoxy polyethylene glycol epoetin beta (0.6 mcg/kg q2w) will be administered using MIRCERA ready-to-use-syringes up to 9 months.

SUMMARY:
This non-interventional, observational study investigates the efficiency, safety and acceptance of MIRCERA in participants, who received erythropoiesis stimulating agent (ESA) using a self-application system. For each participant, the investigator documents 9 months of treatment with Mircera with respect to efficacy, safety and acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Anemia caused by CKD only
* Life expectancy of more than (>) 9 months in the judgment of the attending physician
* Ferritin >200 micrograms per liter (mcg/L) in accordance with the relevant guidelines
* The time point of changing to Mircera was only 3 months ago at the longest

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic kidney disease who received ESA therapy or multidose system before they changed to MIRCERA
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Daun, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- MIRCERA: Participants receiving MIRCERA ready-to-use-syringes (methoxy polyethylene glycol epoetin beta) at the discretion of treating physician were followed for 9 months. The recommended starting dose for MIRCERA in naive participants was 0.6 micrograms per kilogram (mcg/kg) body weight, administered at intervals of 2 weeks. After hemoglobin value reached the target level of 11 grams per deciliter (g/dL), the interval of administration could be adopted to one monthly dose (1.2 mcg/kg body weight)..
Period: Overall Study
Arm/Group | MIRCERA
Started | 240
Completed | 201
Not Completed | 39
Not completed — Death/adverse event | 18
Not completed — Administrative reasons | 3
Not completed — Kidney transplant | 3
Not completed — Lack of Efficacy | 6
Not completed — Consent withdrawn | 7
Not completed — Enrolled but not treated | 2

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who had at least one MIRCERA application.
Groups:
- MIRCERA: Participants receiving MIRCERA ready-to-use-syringes (methoxy polyethylene glycol epoetin beta) at the discretion of treating physician were followed for 9 months. The recommended starting dose for MIRCERA in naive participants was 0.6 mcg/kg body weight, administered at intervals of 2 weeks. After hemoglobin value reached the target level of 11 g/dL, the interval of administration could be adopted to one monthly dose (1.2 mcg/kg body weight).
Arm/Group | MIRCERA
Number analyzed (Participants) | 238
Age, Continuous [Mean (Full Range); unit: years] | 66.8 [24 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 129

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Satisfied With Previous Erythropoiesis Stimulating Agent (ESA) Treatment
Description: Participant satisfaction was measured using 3 categories (1=satisfying, 2=undecided, 3=non- satisfying). Percentage of participants who were satisfied (with a rating of 1 [satisfying]) with previous ESA treatment was reported. For participants who had multiple previous ESA treatments, the latest applied ESA before start of Mircera therapy was considered.
Time Frame: Baseline
Population: Participant Satisfaction Set included all participants who had at least one MIRCERA application, without any major protocol violation and had satisfaction rating documented for previous ESA and MIRCERA.
Measure: Number; unit: percentage of participants
Arm/Group | MIRCERA
Number analyzed (Participants) | 221
percentage of participants | 83.7

2. Primary Outcome: Percentage of Participants Satisfied With the MIRCERA Treatment, Application, Preparation, Storage, and Disposal at Month 1
Description: Participant satisfaction was measured using 3 categories (1=satisfying, 2=undecided, 3=non-satisfying). Percentage of participants who were satisfied (with a rating of 1 [satisfying]) was reported for each of the MIRCERA parameters.
Time Frame: Month 1
Population: Participant Satisfaction Set.
Measure: Number; unit: percentage of participants
Arm/Group | MIRCERA
Number analyzed (Participants) | 221
percentage of participants
  Treatment | 93.7
  Application | 93.7
  Preparation | 95.9
  Storage | 96.8
  Disposal | 92.3

3. Primary Outcome: Percentage of Participants Satisfied With the MIRCERA Treatment, Application, Preparation, Storage, and Disposal at Month 2
Description: as for outcome 2
Time Frame: Month 2
Population: Participant Satisfaction Set. Here number of participants analyzed (N) = participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | MIRCERA
Number analyzed (Participants) | 218
percentage of participants
  Treatment | 93.6
  Application | 92.7
  Preparation | 96.8
  Storage | 96.8
  Disposal | 92.2

4. Primary Outcome: Percentage of Participants Satisfied With the MIRCERA Treatment, Application, Preparation, Storage, and Disposal at Month 3
Description: as for outcome 2
Time Frame: Month 3
Population: Participant Satisfaction Set. Here N = participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | MIRCERA
Number analyzed (Participants) | 218
percentage of participants
  Treatment | 93.9
  Application | 91.5
  Preparation | 94.4
  Storage | 94.4
  Disposal | 89.7

5. Primary Outcome: Percentage of Participants Satisfied With the MIRCERA Treatment, Application, Preparation, Storage, and Disposal at Month 4
Description: as for outcome 2
Time Frame: Month 4
Population: Participant Satisfaction Set. Here N = participants who were available for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | MIRCERA
Number analyzed (Participants) | 218
percentage of participants
  Treatment | 93.8
  Application | 91.4
  Preparation | 94.8
  Storage | 94.8
  Disposal | 90.0

6. Primary Outcome: Percentage of Participants Satisfied With the MIRCERA Treatment, Application, Preparation, Storage, and Disposal at Month 5
Description: as for outcome 2
Time Frame: Month 5
Population: Participant Satisfaction Set. Here N = participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | MIRCERA
Number analyzed (Participants) | 218
percentage of participants
  Treatment | 93.6
  Application | 92.2
  Preparation | 96.1
  Storage | 95.1
  Disposal | 91.2

7. Primary Outcome: Percentage of Participants Satisfied With the MIRCERA Treatment, Application, Preparation, Storage, and Disposal at Month 6
Description: as for outcome 2
Time Frame: Month 6
Population: Participant Satisfaction Set. Here N = participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | MIRCERA
Number analyzed (Participants) | 218
percentage of participants
  Treatment | 93.4
  Application | 92.4
  Preparation | 95.4
  Storage | 95.4
  Disposal | 90.4

8. Primary Outcome: Percentage of Participants Satisfied With the MIRCERA Treatment, Application, Preparation, Storage, and Disposal at Month 7
Description: as for outcome 2
Time Frame: Month 7
Population: Participant Satisfaction Set. Here N = participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | MIRCERA
Number analyzed (Participants) | 218
percentage of participants
  Treatment | 94.8
  Application | 92.7
  Preparation | 94.3
  Storage | 94.8
  Disposal | 89.1

9. Primary Outcome: Percentage of Participants Satisfied With the MIRCERA Treatment, Application, Preparation, Storage, and Disposal at Month 8
Description: as for outcome 2
Time Frame: Month 8
Population: Participant Satisfaction Set. Here N = participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | MIRCERA
Number analyzed (Participants) | 218
percentage of participants
  Treatment | 95.2
  Application | 94.1
  Preparation | 94.1
  Storage | 94.7
  Disposal | 89.3

10. Primary Outcome: Percentage of Participants Satisfied With the MIRCERA Treatment, Application, Preparation, Storage, and Disposal at Month 9
Description: as for outcome 2
Time Frame: Month 9
Population: Participant Satisfaction Set. Here N = participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | MIRCERA
Number analyzed (Participants) | 218
percentage of participants
  Treatment | 94.5
  Application | 94.5
  Preparation | 95.1
  Storage | 94.5
  Disposal | 89.6

11. Secondary Outcome: Change From Baseline in Hemoglobin (Hb) Concentration
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9
Population: Secondary endpoint set included all participants who had at least one MIRCERA application, without any major protocol violation and had at least 6 months documentation and minimum 2 of the 3 visits non-missing Hb and dosing data from Month 7 to 9 visits. N=participants evaluable for this outcome and n=participants evaluable for specified timeframe.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | MIRCERA
Number analyzed (Participants) | 171
g/dL
  Month 1 (n = 34) | 0.02 (0.966)
  Month 2 (n = 166) | -0.03 (1.230)
  Month 3 (n = 163) | -0.26 (1.216)
  Month 4 (n = 165) | -0.36 (1.191)
  Month 5 (n = 161) | -0.31 (1.215)
  Month 6 (n = 152) | -0.34 (1.128)
  Month 7 (n = 171) | -0.38 (1.250)
  Month 8 (n = 159) | -0.31 (1.294)
  Month 9 (n = 86) | -0.29 (1.202)

12. Primary Outcome: Change From Baseline in Pain Sensation Using Visual Analogue Scale
Description: Pain sensation was reported by participants using a visual scale ranging from 0 (no pain) to 10 (strong pain). Pain sensation at baseline referred to pain sensation regarding previous ESA. Change of pain sensation = pain sensation regarding previous ESA (baseline)' minus 'pain sensation regarding MIRCERA (Month 1-9). Positive numbers indicate less pain sensation during MIRCERA application.
Time Frame: Baseline, Months 1-9
Population: Participant Satisfaction Set. Here N = participants who were evaluable for this outcome measure and n = participants evaluable for specified timeframe.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MIRCERA
Number analyzed (Participants) | 214
units on a scale
  Baseline (n =214) | 1.04 (1.205)
  Change at Month 1-9 (n = 178) | 0.33 (1.258)

13. Primary Outcome: Percentage of Participants Who Reported Easement of Therapy With MIRCERA
Time Frame: 9 months
Population: Participant Satisfaction Set.
Measure: Number; unit: percentage of participants
Arm/Group | MIRCERA
Number analyzed (Participants) | 221
percentage of participants | 93.7

14. Primary Outcome: Percentage of Participants Who Continued Treatment After End of Study
Time Frame: End of observation period (Month 9)
Population: Participant Satisfaction Set. Here N = participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | MIRCERA
Number analyzed (Participants) | 142
percentage of participants | 84.5

15. Primary Outcome: Average Monthly Dose of MIRCERA
Time Frame: 9 months
Population: Participant Satisfaction Set. Here N = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | MIRCERA
Number analyzed (Participants) | 142
grams | 144.4 (105.50)

16. Primary Outcome: Number of MIRCERA Dose Adaptations
Time Frame: 9 months
Population: Participant Satisfaction Set. Here N = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: dose adaptations
Arm/Group | MIRCERA
Number analyzed (Participants) | 142
dose adaptations | 3.2 (2.03)

17. Primary Outcome: Mean Monthly Administrations of MIRCERA
Time Frame: 9 months
Population: Efficiency Set included all participants who had at least one MIRCERA application, without any major protocol violation and had prescription and application data available for 2 months before start of MIRCERA and first 2 months of study. Here N = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: MIRCERA administrations per month
Arm/Group | MIRCERA
Number analyzed (Participants) | 142
MIRCERA administrations per month | 1.2 (0.20)

18. Primary Outcome: Percentage of Participants With Pre-Post Shift for Participant Satisfaction With Treatment
Description: Participant satisfaction with treatment was measured using 3 categories (1=satisfying, 2=undecided, 3=non-satisfying). Participant pre-post comparison of satisfaction rating was done by considering the difference of baseline rating (satisfaction rating for previous ESA) and rating at respective visit (satisfaction rating for MIRCERA). Thus, possible results were -2, -1, 0, 1, and 2, with positive values indicating a greater satisfaction with MIRCERA than with the previous ESA (acceptance and preference of MIRCERA over previous ESA). Percentage of participants with each possible result category (-2, -1, 0, 1, 2) is reported at each visit.
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9
Population: Participant Satisfaction Set. Here, n = participants evaluable for specified timeframe.
Measure: Number; unit: percentage of participants
Arm/Group | MIRCERA
Number analyzed (Participants) | 221
percentage of participants
  Month 1: -2 (n=221) | 0.9
  Month 1: -1 (n=221) | 2.7
  Month 1: 0 (n=221) | 81.0
  Month 1: 1 (n=221) | 14.0
  Month 1: 2 (n=221) | 0
  Month 1: No satisfaction rating (n=221) | 1.4
  Month 2: -2 (n=218) | 0.9
  Month 2: -1 (n=218) | 1.4
  Month 2: 0 (n=218) | 79.4
  Month 2: 1 (n=218) | 14.7
  Month 2: 2 (n=218) | 0
  Month 2: No satisfaction rating (n=218) | 3.6
  Month 3: -2 (n=213) | 0.9
  Month 3: -1 (n=213) | 0.9
  Month 3: 0 (n=213) | 80.3
  Month 3: 1 (n=213) | 14.1
  Month 3: 2 (n=213) | 0
  Month 3: No satisfaction rating (n=213) | 3.8
  Month 4: -2 (n=210) | 0
  Month 4: -1 (n=210) | 1.4
  Month 4: 0 (n=210) | 78.6
  Month 4: 1 | 15.2
  Month 4: 2 (n=210) | 0
  Month 4: No satisfaction rating (n=210) | 4.8
  Month 5: -2 (n=204) | 1.0
  Month 5: -1 (n=204) | 1.0
  Month 5: 0 (n=204) | 79.9
  Month 5: 1 (n=204) | 14.2
  Month 5: 2 (n=204) | 0
  Month 5: No satisfaction rating (n=204) | 3.9
  Month 6: -2 (n=197) | 1.0
  Month 6: -1 (n=197) | 1.5
  Month 6: 0 (n=197) | 79.2
  Month 6: 1 (n=197) | 14.2
  Month 6: 2 (n=197) | 0
  Month 6: No satisfaction rating (n=197) | 4.1
  Month 7: -2 (n=192) | 0.5
  Month 7: -1 (n=192) | 0.5
  Month 7: 0 (n=192) | 81.3
  Month 7: 1 (n=192) | 13.5
  Month 7: 2 (n=192) | 0
  Month 7: No satisfaction rating (n=192) | 4.2
  Month 8: -2 (n=187) | 0
  Month 8: -1 (n=187) | 0
  Month 8: 0 (n=187) | 80.7
  Month 8: 1 (n=187) | 14.4
  Month 8: 2 (n=187) | 0
  Month 8: No satisfaction rating (n=187) | 4.9
  Month 9: -2 (n=183) | 0
  Month 9: -1 (n=183) | 0.5
  Month 9: 0 (n=183) | 80.9
  Month 9: 1 (n=183) | 13.7
  Month 9: 2 (n=183) | 0
  Month 9: No satisfaction rating (n=183) | 4.9

ADVERSE EVENTS:
Time Frame: up to the end of study (9 months)
Arm/Group | MIRCERA
Serious Adverse Events (participants affected / at risk) | 27/238
Other Adverse Events (participants affected / at risk) | 9/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MIRCERA (N=238)
Haemoglobin decreased (Investigations) | 11
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 3
Febrile infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Shunt malfunction (Injury, poisoning and procedural complications) | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Hypotension (Vascular disorders) | 1
Extremity necrosis (Vascular disorders) | 1
Diverticulum intestinal haemorrhagic (Vascular disorders) | 1
Bradycardia (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Coronary angioplasty (Surgical and medical procedures) | 1
Arteriovenous shunt operation (Surgical and medical procedures) | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Diverticulitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MIRCERA (N=238)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1
Haematocrit decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.